CLINICAL TRIAL: NCT04998071
Title: Comparison of Analgesic Efficiency in Laparoscopic Percutaneous Extraperitoneal Closure for Pediatric Inguinal Hernia and Hydrocele Provided by Ultrasound Guided Posterior Quadratus Lumborum Block Using Between 0.125% and 0.25% Bupivacaine
Brief Title: Posterior Quadratus Lumborum Block Using 0.125% Versus 0.25% Bupivacaine for Analgesia in Children Undergoing LPEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Sirikit National Institute of Child Health (Other Government)
Responsible Party: Principal Investigator, Kullasate Sakpichaisakul, Queen Sirikit National Institute of Child Health, Queen Sirikit National Institute of Child Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC.015/2564
Record Dates: First submitted 2021-07-09; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROUTINE DRUG - CONCENTRATION QLB (Active Comparator): The patients will receive bilateral posterior quadratus lumborum block using 0.25% bupivacaine 0.4 ml/kg. in each side.
  Interventions: Drug: Bupivacaine hydrochloride
- ALTERNATIVE DRUG - CONCENTRATION QLB (Active Comparator): The patients will receive bilateral posterior quadratus lumborum block using 0.125% bupivacaine 0.4 ml/kg. in each side.
  Interventions: Drug: Bupivacaine hydrochloride

INTERVENTIONS:
Drug: Bupivacaine hydrochloride — Analgesic efficiency comparison between two concentration of bupivacaine hydrochloride using for posterior quadratus lumborum block in LPEC

SUMMARY:
The aim of the present study is to evaluate and compare the analgesic efficiency of the difference concentration between 0.125% and 0.25% bupivacaine provided by ultrasound guided posterior quadratus lumborum block undergoing LPEC in children

DETAILED DESCRIPTION:
Fifty participants both male and female aged from 1 to 6 years old, AGED FROM 1 TO 6 YEARS OLD, ASA class I to II undergoing elective Laparoscopic percutaneous extraperitoneal closure for pediatric inguinal hernia and hydrocele will be randomly divided into two equal groups of twenty five by using computer generated random table.

All received premedication in the form of midazolam 0.1 mcg/kg IV. Perioperative monitoring included continuous ECG, NIBP and pulse oximetry. Baseline reading of these were recorded. General anesthesia will be inducted using thiopental 5 mg/kg then atracurium 0.5 mg/kg to facilitate endotracheal tube intubation and fentanyl 1 mcg/kg. Anesthesia will be maintained using 2% isoflurane with oxygen to air 40:60.

Posterior quadratus lumborum block (The technique which local anesthetic agent is injected at middle thoracolumbar fascia between erector spina muscle and quadratus lumborum muscle) provided by GE, LOGIQe VERSION (12L-RS, LINEAR ARRAY) ultrasound guided and using stimuplex needle 22G-2 inches on both sides under sterile technique in lateral position will be performed in all patients immediately after induction and before starting surgery. patients will be allocated randomly into two equal groups, twenty five in each as the following GROUP 1 will receive 0.25% bupivacaine 0.4 ml/kg. per each side. GROUP 2 will receive 0.125% bupivacaine 0.4 ml/kg. per each side. The patients and parents along with independent anesthesiologist and attending nurses were not aware of group allocation.

The surgical intervention was started not less than 10 minutes after block. Pneumoperitonium pressure was limited not exceed 10 mmHg. After completion of surgery, anesthesia was discontinued and muscle relaxant was reversed as usual. After extubation, the patients will be transfer to PACU.

Postoperative pain will be assessed by attending nurses, using CHEOPs SCORE. Acetaminophen 10 mg/kg. orally will be given as rescue analgesia for patient with CHEOPs SCORE more than 6. Parameters will be assessed

Intraoperative measurements:

1. Hemodynamic parameters: HR and MAP were recorded before, immediately and every 5 minutes after induction of anesthesia until the end of the operation.
2. Analgesic requirement: All through the procedure (By measure analgesic need intraoperative in the form of fentanyl 0.5 mcg/kg) In case of increase in intraoperative MAP or HR of more than 20% from baseline.
3. Incidence of complications: In the form of hypotension, hematoma, intraabdominal organ injury LAST.

Postoperative measurements:

1. Quality of analgesia: Assessed immediately postoperatively every 30 minutes in the PACU and then at 4, 8, 12 hours at ward using CHEOPs SCORE and 24 hours postoperatively using PARENT'S POSTOPERATIVE PAIN MEASUREMENT(PPPM).
2. Incidence of complications: In the form assessment of intensity of motor block by using MODIFIED BROMAGE SCORE, vomiting and hemodynamic instability.
3. Others: In the form of parent's satisfaction of analgesia and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for laparoscopic percutaneous extraperitoneal closure(LPEC) for pediatric inguinal hernia and hydrocele
* ASA I-II physical status patients
* Complete inform consent for intervention

Exclusion Criteria:

* Contraindication for regional anesthesia
* Sensitive to local anesthetic agent, opioid or acetaminophen
* Previous history of abdominal surgery
* History of neuromuscular disease
* G6PD deficiency

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of postoperative analgesia | 24 hours after surgery
  Postoperative pain score as CHEOPs SCORE

SECONDARY OUTCOMES:
Incidence of complications | 12 hours after surgery
  Intensity of motor block by using MODIFIED BROMAGE SCORE, vomiting and hemodynamic instability

CONTACTS AND LOCATIONS:
Overall Officials: SUWITCHA TAMRONGCHOTE, MD, Principal Investigator — Queen Sirikit National Institute of Child Health (QSNICH)
Locations (1):
- Queen Sirikit National Institute of Child Health, Ratchathewi, Bangkok, Thailand